CLINICAL TRIAL: NCT01042678
Title: A Phase I/II, Open-label, Single Ascending Dose Study Evaluating the Safety, Preliminary Efficacy, and Pharmacokinetics of Intravitreal MP0112 in Patients With Diabetic Macular Edema (DME)
Brief Title: Study of MP0112 Intravitreal Injection in Patients With Diabetic Macular Edema
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a company decision.
Sponsor: Allergan (Industry)
Collaborators: Molecular Partners AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP0112-CP02
Record Dates: First submitted 2010-01-01; First posted 2010-01-05 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — MP0112

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- MP0112 (0.04 mg) (Experimental): Single 0.04 mg intravitreal injection of MP0112 in the study eye.
  Interventions: Biological: MP0112
- MP0112 (0.15 mg) (Experimental): Single 0.15 mg intravitreal injection of MP0112 in the study eye.
  Interventions: Biological: MP0112
- MP0112 (0.4 mg) (Experimental): Single 0.4 mg intravitreal injection of MP0112 in the study eye.
  Interventions: Biological: MP0112
- MP0112 (1.0 mg) (Experimental): Single 1.0 mg intravitreal injection of MP0112 in the study eye.
  Interventions: Biological: MP0112
- MP0112 (2.0 mg) (Experimental): Single 2.0 mg intravitreal injection of MP0112 in the study eye.
  Interventions: Biological: MP0112
- MP0112 (3.6 mg) (Experimental): Single 3.6 mg intravitreal injection of MP0112 in the study eye.
  Interventions: Biological: MP0112

INTERVENTIONS:
Biological: MP0112 — Single intravitreal injection of MP0112 in the study eye

SUMMARY:
The purpose of this study is to assess the safety and tolerability of MP0112 (a novel, potentially long acting VEGF inhibitor) in patients with diabetic retinal edema.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 years or older
* Macular edema due to diabetic retinopathy
* Best-corrected visual acuity in the study eye of 20/40 to 20/400
* Central subfield thickness ≥ 250 microns by OCT
* Females of childbearing potential must have a negative serum pregnancy test at Screening
* Male subjects must or be: 1) surgically sterilized for at least 6 months, or 2) use an appropriate method of barrier contraception (e.g., condoms with spermicide) and advise any sexual partner of child-bearing potential that she must also use a reliable method of contraception (e.g., hormonal contraceptive, intrauterine device, diaphragm with spermicide) during the study and for 30 days from study drug administration.
* Ability to understand the nature of the study and give written informed consent
* Willing, committed, and able to return for ALL clinic visits and complete all study-related procedures

Exclusion Criteria:

* Any indication of irreversible vision loss such as significant atrophy, scarring, fibrosis, or hyperpigmentation in the fovea
* Presence of significant ocular abnormalities in the study eye that prevent retinal assessment, including media opacities, cataract, or inadequate papillary dilation
* Presence of vision loss from another ocular disease other than DME
* History of any intraocular surgery within 3 months of Baseline
* History of intraocular injection of anti-VEGF agent or steroids within 3 months of Baseline
* History of laser photocoagulation for macular edema within 4 months prior to Baseline
* Uncontrolled hypertension > 140 systolic or > 95 diastolic
* HbA1C ≥ 12%
* Creatinine: > 1.5 x upper limit of normal (ULN)
* Alanine transaminase (ALT), aspartate transaminase (AST), and gamma-glutamyl transferase (GGT): > ULN
* White blood cells (WBC), hematocrit, and platelets: < lower limit of normal (LLN)
* Heart rate < 60 beats per minute (bpm) or history of clinically significant bradycardia
* History of human immunodeficiency virus (HIV), chronic hepatitis B, or chronic hepatitis C infections
* Subjects with infections requiring hospitalization and/or antibiotic treatment 14 days prior to Baseline
* Subjects with any medical condition that in the judgment of the investigator could poise unacceptable risk to the subject or compromise interpretation of the data to be collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Wilmer Eye Institute, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Research Center, Austin, Texas
  - Retina Consultants of Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg) | MP0112 (1.0 mg) | MP0112 (2.0 mg) | MP0112 (3.6 mg)
Started | 6 | 6 | 6 | 0 | 0 | 0
Completed | 5 | 6 | 6 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (8.4) | 67.5 (9.9) | 64.2 (10.3) | 64.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 4 | 3 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Safety and tolerability was assessed by vital signs, clinical laboratory evaluations, ophthalmological examinations, intraocular pressure, the presence of anti-drug antibodies and the collection of adverse events. An adverse event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events.
Time Frame: 16 weeks
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg)
Number analyzed (Participants) | 6 | 6 | 6
Participants
  Adverse Events (AEs) | 3 | 6 | 6
  Serious Adverse Events | 0 | 1 | 0
  Ophthalmic AEs in the Study Eye | 3 | 5 | 5
  Ophthalmic AEs in the Fellow Eye | 1 | 3 | 5

2. Secondary Outcome: Best-Corrected Visual Acuity (BCVA)
Description: BCVA was measured using an eye chart and was reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye at Baseline and Week 16. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the letters read correctly on the eye chart the better the vision.
Time Frame: Baseline, Week 16
Population: All treated participants with data for a given time point were included for analysis.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg)
Number analyzed (Participants) | 6 | 6 | 6
Letters
  Baseline (n=5,4,5) | 56.2 (9.8) | 59.0 (4.8) | 59.6 (17.1)
  Week 16 (n=5,6,5) | 66.8 (12.9) | 55.5 (10.0) | 66.0 (17.5)

3. Secondary Outcome: Change From Baseline in Foveal Thickness as Measured by Optical Coherence Tomography (OCT)
Description: Optical Coherence Tomography (OCT), a laser based non-invasive diagnostic system providing high-resolution imaging sections of the fovea (part of the retina), was performed in the study eye after pupil dilation at Baseline and Week 16. A negative change from Baseline indicated improvement (less foveal thickness).
Time Frame: Baseline, Week 16
Population: All treated participants.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg)
Number analyzed (Participants) | 6 | 6 | 6
microns
  Baseline | 390.5 (104.3) | 514.3 (146.0) | 402.0 (98.8)
  Change from Baseline at Week 16 (n=5,6,5) | -8.8 (78.4) | -57.8 (170.3) | -29.2 (96.0)

4. Secondary Outcome: Serum Levels of MP0112
Description: Blood samples were collected Pre-treatment (Baseline), Day 1 and 3, Weeks 1, 4, 12, 16. Serum samples (liquid portion of the blood after cells and clotting factors were removed) were sent to a laboratory for analysis. Levels of MP0112 were determined using an enzyme-linked immunosorbent assay.
Time Frame: 16 Weeks
Population: All treated participants.
Measure: Median (Full Range); unit: Nanomolar (nM)
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg)
Number analyzed (Participants) | 6 | 6 | 6
Nanomolar (nM) | NA [NA to NA] — Result below Lower Limit of Quantification of the Assay =0.3 nM. | NA [NA to NA] — Result below Lower Limit of Quantification of the Assay=0.3 nM. | NA [NA to NA] — Result below Lower Limit of Quantification of the Assay=0.3 nM.

5. Secondary Outcome: Aqueous Humor Levels of MP0112
Description: Aqueous humor (the thin, watery fluid in the eye) samples were collected from anterior chamber taps and were sent to a laboratory for analysis. Levels of MP0112 were determined using an enzyme-linked immunosorbent assay.
Time Frame: 1 Week
Population: All treated participants who consented to participate.
Measure: Median (Full Range); unit: nM
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg)
Number analyzed (Participants) | 3 | 3 | 4
nM | 14 [13 to 26] | 106 [26 to 270] | 555 [230 to 622]

6. Secondary Outcome: Number of Participants With Positive Binding Anti-MP0112 Antibodies
Description: Blood samples were collected Pre-treatment (Baseline) and Weeks 4, 8 and 12. Samples were analyzed for Anti-MP0112 antibodies using an enzyme-linked immunosorbent assay.
Time Frame: 12 weeks
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg)
Number analyzed (Participants) | 6 | 6 | 6
Participants | 0 | 0 | 3

ADVERSE EVENTS:
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg)
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP0112 (0.04 mg) (N=6) | MP0112 (0.15 mg) (N=6) | MP0112 (0.4 mg) (N=6)
Chest pain (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MP0112 (0.04 mg) (N=6) | MP0112 (0.15 mg) (N=6) | MP0112 (0.4 mg) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 2 | 2 | 3
Foreign body sensation in eyes (Eye disorders) | 3 | 2 | 1
Anterior chamber flare (Eye disorders) | 0 | 0 | 5
Eye pain (Eye disorders) | 1 | 2 | 2
Iritis (Eye disorders) | 0 | 2 | 2
Conjunctival hyperaemia (Eye disorders) | 1 | 1 | 1
Eye irritation (Eye disorders) | 1 | 1 | 1
Anterior chamber cell (Eye disorders) | 0 | 0 | 2
Blepharitis (Eye disorders) | 1 | 0 | 1
Conjunctival oedema (Eye disorders) | 0 | 2 | 0
Photophobia (Eye disorders) | 0 | 2 | 0
Retinal exudates (Eye disorders) | 1 | 0 | 1
Vitreal cells (Eye disorders) | 0 | 0 | 2
Vitreous floaters (Eye disorders) | 0 | 1 | 1
Vitritis (Eye disorders) | 0 | 2 | 0
Diabetic retinal oedema (Eye disorders) | 0 | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0 | 0
Iris adhesions (Eye disorders) | 0 | 1 | 0
Iris atrophy (Eye disorders) | 0 | 1 | 0
Lenticular pigmentation (Eye disorders) | 0 | 1 | 0
Macular oedema (Eye disorders) | 0 | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 0 | 1
Punctate keratitis (Eye disorders) | 0 | 0 | 1
Retinal cyst (Eye disorders) | 1 | 0 | 0
Retinal ischaemia (Eye disorders) | 0 | 1 | 0
Retinal neovascularisation (Eye disorders) | 0 | 1 | 0
Retinal pigment epitheliopathy (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 1 | 0
Vitreous fibrin (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 1 | 0
Paracentesis eye (Investigations) | 0 | 1 | 0
Protein urine present (Investigations) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.